CLINICAL TRIAL: NCT00181740
Title: A Pilot Study of Concerta Treatment in Adults With Attention Deficit Hyperactivity Disorder Not Otherwise Specified
Brief Title: Concerta Treatment in Adults With ADHD NOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc. (Industry)
Responsible Party: Joseph Biederman, MD, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003-P-001355
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2010-07-23 (Estimated); Status verified 2010-07

CONDITIONS: ADHD NOS
Keywords: ADHD NOS; Adults; Concerta; Open-Label
MeSH Terms: interventions — Atomoxetine Hydrochloride

INTERVENTIONS:
Drug: atomoxetine (Strattera)

SUMMARY:
This will be an open label pilot study of Concerta in the treatment of adults with the diagnosis of Attention Deficit Hyperactivity Disorder Not Otherwise Specified (ADHD NOS). We hypothesize ADHD symptomatology in adults with ADHD NOS will be responsive to Concerta treatment in the short term and Concerta-associated response of ADHD symptomatology in adults with ADHD NOS will be sustained over the medium term.

DETAILED DESCRIPTION:
Concerta is a stimulant medication approved for the treatment of ADHD in children. We propose to study the safety and efficacy of Concerta therapy in adults with ADHD NOS. Adult ADHD NOS is operationalized by either

* An adult satisfying current diagnostic criteria for ADHD but with insufficient number of childhood symptoms to fulfill the required diagnostic threshold for this disorder set forth in DSM-IV
* An adult who has five current symptoms of inattention and/or five current symptoms of impulsivity/hyperactivity, but does not meet the full diagnosis criteria of six current symptoms within one of these categories.

Our hypotheses will be examined in two phases of an open label, pilot study. Phase I of the study consists of a six-week acute effectiveness trial. Phase II consists of continuation for responders in which subjects who respond in Phase I will be re-assessed every four weeks for six months. Effectiveness will be measured by improvements in clinician-rated scales, including: ADHD Symptom Checklist, Clinical Global Impression: ADHD, and Global Assessment of Functioning.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female outpatients older than 18 and younger than 55 years of age.
2. Subjects with the diagnosis of Attention Deficit Hyperactivity Disorder Not Otherwise Specified (ADHD NOS), by DSM-IV, as manifested in clinical evaluation and confirmed by structured interview. This is operationalized by either

   * Having at least 5 out of 9 current DSM-IV items of either inattention or hyperactivity/impulsivity but < 5 items from either list in childhood
   * Having 5 out of 9 current DSM-IV items of either inattention or hyperactivity/impulsivity, but not having the 6 current symptoms in either category. This second category will be included independent of the presence or absence of ADHD symptoms in childhood.
3. Subjects will have a current Clinical Global Impression: ADHD score of 4 (moderately ill) or higher illness severity.
4. Patients with past history of depression, bipolar disorder, anxiety disorder (including OCD) without current disorder for > 3 months as ascertained through structured diagnostic interview and clinical exam.
5. Subjects treated for anxiety disorders and depression who are on a stable medication regimen for at least three months, and who have a disorder specific CGI-severity score ≤ 3 (mildly ill) and who have a score on the Hamilton-Depression and Hamilton-anxiety rating scale below 15 (mild range) will be included in the study.
6. Subjects with a past history of tics but tic free for > 1 year.
7. Subjects with past history of substance use disorders, but substance free for > 6 months.
8. Subjects receiving non-MAOI antidepressants (e.g., SSRI's, bupropion, venlafaxine), or benzodiazepines who have been on a stable regimen for > 3 months for any of the conditions listed above. Subjects taking SSRIs will be allowed into the study for the following reasons:

   * SSRIs are not known to interact with methylphenidate
   * Methylphenidate metabolism does not involve the hepatic P450 enzymatic system
   * SSRIs have extremely wide margins of safety
   * SSRIs and methylphenidate are combined routinely in clinical practice.
9. Subjects with mild cases of asthma and allergy will not be excluded.
10. Subjects with acid reflux syndrome will not be excluded.
11. Subjects with hypercholesterolemia will not be excluded.

Exclusion Criteria:

1. Any clinically unstable psychiatric conditions including the following: acute psychosis, acute panic, acute OCD, acute mania, acute suicidality, bipolar disorder, acute substance use disorders (alcohol or drugs), acute OCD, sociopathy, criminality.
2. Any metabolic, neurological, hepatic, renal, cardiovascular, hematological, opthalmic, or endocrine disease.
3. Clinically significant abnormal baseline laboratory values which include the following:

   * Values larger than 20% above the upper range of the laboratory standard of a basic metabolic screen.
   * Exclusionary blood pressure parameters will include any values above 140 (systolic) and 90 (diastolic).
   * Exclusionary ECG parameters will include a QTC> 460msec, QRS>120 msec, and PR>200 msec. Subjects having ECG evidence of ischemia or arrhythmia as reviewed by an independent cardiologist.
4. Mental retardation (I.Q. <75).
5. Organic brain disorders.
6. Seizures or tics in the last year.
7. Subjects with a family history or diagnosis of Tourette's syndrome.
8. Subjects who are being treated with monoamine oxidase inhibitors, or have stopped treatment of monoamine oxidase inhibitors for less than 14 days prior to baseline visit.
9. Subjects taking coumadin anticoagulants, anticonvulsants, or tricyclic antidepressants.
10. Pregnant or nursing females.
11. Subjects with current adequate treatment for ADHD or a history of a previous adequate trial of Concerta.
12. Non English speaking subjects will not be allowed into the study for the following reasons:

    * The assessment instruments are not available and have not been adequately standardized in other languages
    * Our clinical trials facility is located in Cambridge and not in the MGH main campus without the availability of translators
    * Psychiatric questionnaires and evaluations are taxing and adding the complexity of a translator has the potential to make the patient experience even more exhausting.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30
Dates: Start 2003-12; Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
improvement of ADHD symptoms as related by scores on the
ADHD Symptom Checklist
Clinical Global Impression: ADHD
Global Assessment of Functioning

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Biederman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Cambridge, Massachusetts, United States